CLINICAL TRIAL: NCT06354673
Title: Stellate Ganglion Block Combined With Dexmedetomidine or Subanesthetic Ketamine Infusion for Treatment of Neurostorm After Traumatic Brain Injury in Critically Ill Patients: A Randomized Clinical Study.
Brief Title: Stellate Ganglion Block Combined With Dexmedetomidine or Subanesthetic Ketamine Infusion for Treatment of Neurostorm.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 278/1-April-2024
Record Dates: First submitted 2024-04-04; First posted 2024-04-09 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2024-04

CONDITIONS: Paroxysmal Sympathetic Hyperactivity
MeSH Terms: interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SD group (Experimental): Stellate ganglion block and 1 ug/kg/h intravenous Dexmedetomidine infusion
  Interventions: Procedure: Stellate ganglion block; Drug: Dexmedetomidine
- SK group (Experimental): Stellate ganglion block and 0.5 mg/kg/h intravenous ketamine infusion.
  Interventions: Procedure: Stellate ganglion block; Drug: Ketamine

INTERVENTIONS:
Procedure: Stellate ganglion block — Sympathectomy by using combination of regional nerve block and systemic drugs
Drug: Dexmedetomidine — intravenous Dexmedetomidine infusion
  Other Names: Precedex
  Arms: SD group
Drug: Ketamine — intravenous ketamine infusion
  Arms: SK group

SUMMARY:
Neurostorming is a sudden and exaggerated stress response as a result of damage to the brain. With appropriate treatment and time, there is hope for individuals to overcome storming, regain consciousness, and work towards successfully recovering from brain injury. Most treatments for neurostorming involve the use of medications only such as dexmedetomidine, opioids, gabapentin and propofol to address secondary complications like high blood pressure and fever. These medications focus on slowing the body's stress response or relaxing the body. Stellate ganglion block (SGB) is a promising therapy for paroxysmal sympathetic hyperactivity (PSH), overcoming the limitations of systemic medications and may serve to recalibrate aberrant autonomic states. Ketamine is a potent dissociative agent which has sedative, analgesic and anesthetic properties beside its sympathomimetic effect. Its combination with stellate ganglion block is to oppose its sympathomimetic effect. Dexmedetomidine has analgesic and sedative effect which inhibits the sympathetic nerve activity through its action on the α2 receptor in the spinal cord. Hypothesis: Null hypothesis: There is no difference between the effects of stellate ganglion block combined with dexmedetomidine or subanesthetic ketamine infusion for treatment of neurostorm after traumatic brain injury in critically ill patients.Alternative hypothesis: There is a difference between the effects of stellate ganglion block combined with dexmedetomidine or subanesthetic ketamine infusion for treatment of neurostorm after traumatic brain injury in critically ill patients.which has sedative, analgesic and anesthetic properties beside its sympathomimetic effect. Aim of the work is achievement of effective treatment for the neurostorm after traumatic brain injury in critically ill patients with better outcomes and decrease intensive care unit (ICU) stay.

DETAILED DESCRIPTION:
PATIENTS AND METHODS

I. Technical Design:

1. Site of study:

   This study will be carried out in the emergency intensive Care unit (ICU) of Zagazig University Hospitals within 6 months.
2. Sample size:

   The sample size was collected using G power version 3.1.9.7 according to the following expected moderate effect size between stellate ganglion plus dexmedetomidine group (SD group) and stellate ganglion block plus ketamine group (SK group) (d=0.5) CI 95% and power 80% the sample size was calculated to be 102,51 in each group.
3. Patients included in this study:

   * Inclusion criteria:

     1. Written informed consent from 1st degree relative.
     2. Physical ASA status I & II.
     3. BMI less than or equal 35.
     4. Traumatic brain injury patients.
     5. Age: ≥18 years old.
     6. Sex: both sexes.
     7. Paroxysmal sympathetic hyperactivity will be diagnosed on the basis of diagnostic criteria proposed by Blackman et al.(2), The signs of PAID syndrome include: (1) Severe brain injury (Rancho Los Amigos level IV), (2) temperature of at least 38.5°C, (3) pulse of at least 130 beats/min, (4) respiratory rate of at least 140 breaths/min, (5) agitation, (6) diaphoresis, and (7) dystonia (i.e. rigidity or decerebrate posturing). The duration is at least1 cycle/day for at least 3 days.
   * Exclusion criteria:

     1. Known hypersensitivity to study drugs.
     2. Patients with primary brain stem injury or brain stem hemorrhage
     3. Severe systemic organ diseases.
     4. GCS score =3 points
     5. Patients complicated with severe coagulation abnormalities, hemorrhagic shock, multiple organ failure.
     6. Patients with a history of cerebral hemorrhage or cerebral infarction within the past three months.
     7. Patients complicated with a history of end stage malignancy.
     8. Patients complicated with a history of uncontrolled epilepsy.

Withdrawal criteria:

The patient has the right to withdraw from the study at any time without any negative consequence on their medical treatment plan.

II. Operational Design:

1. Type of study:

   Double-blinded randomized clinical trial.
2. Parameters of the study will include:

All patients suspected of having PSH will underwent detailed clinical history and physical examination. Hemodynamics monitoring including heart rate and mean arterial pressure (MAP) also temperature monitoring will be done as base line before the block and after stellate ganglion block every one hour over 24 hours until remission (till return to normal values for age and sex). These patients will be also subjected to routine hematological investigations including, complete blood count, kidney and liver function test, coagulation profile, urine analysis for myoglobinuria and thyroid profile. septic screening including, blood, urine, tracheal aspirate and sputum culture and radiological assessment by using chest x-ray.

All patients developing PSH will be randomly allocated by using computerized generated randomization table into two groups:

SD group: Stellate ganglion block and 1 ug/kg/h intravenous Dexmedetomidine infusion.

SK group: Stellate ganglion block and 0.5 mg/kg/h intravenous ketamine infusion.

Stellate ganglion block :

Patients will undergo an ultrasonography-guided SGB at bedside under standard American Society of Anesthesiologists monitoring standards. The patient will be placed in supine position with the head turn to the opposite side. The anterior and lateral parts of the neck will be prepped with chlorhexidine, and a linear (13-6 MHz) ultrasound probe will be applied to the anterolateral neck at the cricoid cartilage level to identify the transverse process of C6 and C7, anterior tubercle of C6 (Chassaignac tubercle), longus colli muscle and surrounding neurovascular structure. The needle will be advanced with an in-plane technique and aimed to deposit the local anesthetics medial to the Chassaignac tubercle and anterior to pre-vertebral fascia of longus colli muscle. After that, a catheter will be advanced through the needle and secured in place. After aspiration, 10 ml of bupivacaine 0.25% solution will be injected through the catheter and repeated every 48 hours till time of remission.

a. Data to be measured:

1. Demographic data including, age, sex, BMI, ASA classification.
2. Hemodynamics including, MAP and heart rate and temperature measurement as base line before stellate ganglion block, after stellate ganglion block and furtherly every hour over 24 hours till time of remission (return to normal value for age and sex).
3. Remission time of paroxysmal hypertension (min): time from the start of treatment till return to normal blood pressure).
4. Remission time of paroxysmal tachycardia (min): time from the start of treatment till return to normal heart rate).
5. Remission time of paroxysmal hypermyotonia (day): the criteria of muscle hyperactivity is the rigid posture or sever dystonia (i.e. rigidity or decerebrate posturing).
6. Remission time of decrease respiratory rate below 25 breath/min (min): time from the start of treatment till time of decrease respiratory rate below 25 breath/min.
7. Changes in glascow coma scale score (GSC) from admission to ICU till discharge: GSC will be evaluated once daily.
8. Duration of ICU stay (days): the duration from the admission till discharge from ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from 1st degree relative.
2. Physical ASA status I & II.
3. BMI less than or equal 35.
4. Traumatic brain injury patients.
5. Age: ≥18 years old.
6. Sex: both sexes.
7. Paroxysmal sympathetic hyperactivity will be diagnosed on the basis of diagnostic criteria proposed by Blackman et al.(2), The signs of PAID syndrome include: (1) Severe brain injury (Rancho Los Amigos level IV), (2) temperature of at least 38.5°C, (3) pulse of at least 130 beats/min, (4) respiratory rate of at least 140 breaths/min, (5) agitation, (6) diaphoresis, and (7) dystonia (i.e. rigidity or decerebrate posturing). The duration is at least 1 cycle/day for at least 3 days

Exclusion Criteria:

* 1) Known hypersensitivity to study drugs. 2) Patients with primary brain stem injury or brain stem hemorrhage 3) Severe systemic organ diseases. 4) GCS score =3 points 5) Patients complicated with severe coagulation abnormalities, hemorrhagic shock, multiple organ failure.

  6) Patients with a history of cerebral hemorrhage or cerebral infarction within the past 3 months. 7) Patients complicated with a history of end stage malignancy.

  8) Patients complicated with a history of uncontrolled epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
To compare the time of remission of neurostorm symptoms | 6 months
  Elevated blood pressure,tachycardia, fever and tachypenea of traumatic brain injury (TBI) between the stellate ganglion block combined with either dexmedetomidine or subanesthetic keyamine infusion
To assess effect of stellate ganglion block combined with either dexmedetomidine or subanesthetic ketamine infusion on changes in glascow coma scale score. | 6 months
  Daily evaluation of glascow coma scale score in which the lowest score is 3 ( indicates poor prognosis) and the highest is 15 (indicates the best prognosis)

SECONDARY OUTCOMES:
▪ To measure the duration of intensive care unit (ICU) stay. | 6months
  Time of patient stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Eslam S. Almaghawry Mohamed, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig university, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meyfroidt G, Baguley IJ, Menon DK. Paroxysmal sympathetic hyperactivity: the storm after acute brain injury. Lancet Neurol. 2017 Sep;16(9):721-729. doi: 10.1016/S1474-4422(17)30259-4. PMID 28816118
- [Background] Blackman JA, Patrick PD, Buck ML, Rust RS Jr. Paroxysmal autonomic instability with dystonia after brain injury. Arch Neurol. 2004 Mar;61(3):321-8. doi: 10.1001/archneur.61.3.321. PMID 15023807
- [Background] Doi S, Cho N, Obara T. Stellate ganglion block increases blood flow in the anastomotic artery after superficial temporal artery-middle cerebral artery bypass. Br J Anaesth. 2016 Sep;117(3):395-6. doi: 10.1093/bja/aew230. No abstract available. PMID 27543535
- [Background] Jain V, Rath GP, Dash HH, Bithal PK, Chouhan RS, Suri A. Stellate ganglion block for treatment of cerebral vasospasm in patients with aneurysmal subarachnoid hemorrhage - A preliminary study. J Anaesthesiol Clin Pharmacol. 2011 Oct;27(4):516-21. doi: 10.4103/0970-9185.86598. PMID 22096287
- [Background] Lipov E, Sethi Z, Nandra G, Frueh C. Efficacy of combined subanesthetic ketamine infusion and cervical sympathetic blockade as a symptomatic treatment of PTSD/TBI in a special forces patient with a 1-year follow-up: A case report. Heliyon. 2023 Mar 27;9(4):e14891. doi: 10.1016/j.heliyon.2023.e14891. eCollection 2023 Apr. PMID 37089345
- [Background] Peters AJ, Villasana LE, Schnell E. Ketamine Alters Hippocampal Cell Proliferation and Improves Learning in Mice after Traumatic Brain Injury. Anesthesiology. 2018 Aug;129(2):278-295. doi: 10.1097/ALN.0000000000002197. PMID 29734230
- [Background] Browne CA, Wulf HA, Jacobson ML, Oyola MG, Wu TJ, Lucki I. Long-term increase in sensitivity to ketamine's behavioral effects in mice exposed to mild blast induced traumatic brain injury. Exp Neurol. 2022 Apr;350:113963. doi: 10.1016/j.expneurol.2021.113963. Epub 2021 Dec 28. PMID 34968423